CLINICAL TRIAL: NCT01527916
Title: A Randomized, Double-Blind, Placebo and Active-Controlled Study to Evaluate the Efficacy and Safety of ABT-126 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Evaluate the Efficacy and Safety of ABT-126 in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M10-985; 2011-002004-32 (EudraCT Number)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; ABT-126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- sugar pill (Placebo Comparator)
  Interventions: Drug: placebo
- donepezil (Active Comparator)
  Interventions: Drug: donepezil
- ABT-126 Low Dose (Experimental): low dose
  Interventions: Drug: ABT-126
- ABT-126 Middle Dose (Experimental): middle dose
  Interventions: Drug: ABT-126
- ABT-126 high dose (Experimental): high dose
  Interventions: Drug: ABT-126

INTERVENTIONS:
Drug: placebo — Placebo Comparator
  Arms: sugar pill
Drug: donepezil — Active Comparator
  Arms: donepezil
Drug: ABT-126 — low dose, middle dose, high dose
  Arms: ABT-126 Low Dose; ABT-126 Middle Dose; ABT-126 high dose

SUMMARY:
This is an efficacy and safety study evaluating a new treatment for subjects with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the efficacy and safety of ABT-126 in approximately 410 adults with mild to moderate Alzheimer's disease. Subjects will be randomized to one of 5 treatment groups (ABT-126, donepezil or placebo) for a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The subject and caregiver must voluntarily sign and date an informed consent. If the subject does not have the capacity to provide informed consent, full informed consent must be obtained from the subject's representative and assent must be obtained from the subject.
* The subject is a male or female between the ages of 55 and 90 years, inclusive, at Screening Visit 1.
* The subject meets the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable Alzheimer's disease.
* The subject has a Mini-Mental Status Examination (MMSE) total score of 10 to 24, inclusive, at Screening Visit 1.
* The subject has a Cornell Scale for Depression in Dementia (CSDD) score ≤ 10 at Screening Visit 1.
* The subject has a Modified Hachinski Ischemic Scale (MHIS) score of ≤ 4 at Screening Visit 1.
* With the exception of a diagnosis of mild to moderate AD and the presence of stable medical conditions, the subject is in general good health, based upon the results of medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).
* The subject has an identified, reliable caregiver who will provide support and ensure compliance with the study medication and procedures, and provide accurate information about the subject's status during the study.

Exclusion Criteria:

* The subject is currently taking or has taken a medication for the treatment of Alzheimer's disease or dementia within 60 days prior to Screening Visit 1, or is participating in cognitive therapy for the treatment of Alzheimer's disease or dementia.
* The subject has clinically significant abnormal laboratory values at Screening Visit 1 as determined by the investigator.
* The subject has a history of any significant neurologic disease other than Alzheimer's disease including Parkinson's disease, multi-infarct or vascular dementia, Huntington's disease, normal pressure hydrocephalus, progressive supranuclear palsy, multiple sclerosis, any seizures, mental retardation or a history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
* In the opinion of the investigator, the subject has any clinically significant uncontrolled medical or psychiatric illness.
* The subject has a known hypersensitivity or intolerance to donepezil that lead to discontinuation or a known reported history of donepezil treatment failure.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - cognitive subscale | Measurements up through 24 weeks

SECONDARY OUTCOMES:
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | Measurements up through 24 weeks
  Caregiver-based assessment of activities of daily living
Mini Mental Status Exam (MMSE) | Measurements up through 24 weeks
  Questionnaire which provides a quantitative measure of cognition
DEMentia Quality of Life (DEMQOL) | Measurements up through 24 weeks
  Health-related quality of life measurement tool
Clinician Interview-Based Impression of Change - plus (CIBIC-plus) | Measurements up through 24 weeks
  Measures a global impression of change in severity of dementia
Neuropsychiatry Inventory (NPI) | Measurements up through 24 weeks
  Assesses the presence of psychopathology in subjects with Alzheimer's disease and other dementias
Partner-Patient Questionnaire for Shared Activities (PPQSA) | Measurements up through 24 weeks
  Measures the extent to which mood and mental state interferes with the patient-partner relationship
Resource Use in Dementia (RUD-Lite) | Measurements up through 24 weeks
  Brief measurement tool for resource utilization
EuroQol-5D Questionnaires | Measurements up through 24 weeks
  Assesses patient's mobility, self-care, usual activity, pain/discomfort and anxiety/depression
Wechsler Memory Scale-III (WMS-III) Working Memory Index | Measurements up through 24 weeks
  Assesses working memory

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD, Study Director — AbbVie
Locations (33):
- United States (8):
  - Site Reference ID/Investigator# 56503, Delray Beach, Florida
  - Site Reference ID/Investigator# 56518, Tampa, Florida
  - Site Reference ID/Investigator# 56514, West Palm Beach, Florida
  - Site Reference ID/Investigator# 62611, Elk Grove Village, Illinois
  - Site Reference ID/Investigator# 56506, Staten Island, New York
  - Site Reference ID/Investigator# 82994, Jenkintown, Pennsylvania
  - Site Reference ID/Investigator# 77636, Wichita Falls, Texas
  - Site Reference ID/Investigator# 56504, Bennington, Vermont
- Poland (3):
  - Site Reference ID/Investigator# 62565, Gdynia
  - Site Reference ID/Investigator# 62563, Poznan
  - Site Reference ID/Investigator# 62562, Szczecin
- Russia (11):
  - Site Reference ID/Investigator# 60945, Kazan'
  - Site Reference ID/Investigator# 60955, Kazan'
  - Site Reference ID/Investigator# 60954, Kirov
  - Site Reference ID/Investigator# 60951, Moscow
  - Site Reference ID/Investigator# 60959, Moscow
  - Site Reference ID/Investigator# 60946, Novosibirsk
  - Site Reference ID/Investigator# 60947, Saint Petersburg
  - Site Reference ID/Investigator# 60958, Saint Petersburg
  - Site Reference ID/Investigator# 60949, Saint Petersburg
  - Site Reference ID/Investigator# 60952, Saint Petersburg
  - Site Reference ID/Investigator# 60950, Saratov
- South Africa (4):
  - Site Reference ID/Investigator# 60911, Belville
  - Site Reference ID/Investigator# 76073, Cape Town
  - Site Reference ID/Investigator# 60912, George
  - Site Reference ID/Investigator# 60910, Johannesburg
- Ukraine (3):
  - Site Reference ID/Investigator# 60909, Donetsk
  - Site Reference ID/Investigator# 60906, Kiev
  - Site Reference ID/Investigator# 60905, Poltava
- United Kingdom (4):
  - Site Reference ID/Investigator# 60960, Bath
  - Site Reference ID/Investigator# 60963, Blackburn
  - Site Reference ID/Investigator# 60962, Glasgow
  - Site Reference ID/Investigator# 60961, London

REFERENCES:
- [Derived] Gault LM, Lenz RA, Ritchie CW, Meier A, Othman AA, Tang Q, Berry S, Pritchett Y, Robieson WZ. ABT-126 monotherapy in mild-to-moderate Alzheimer's dementia: randomized double-blind, placebo and active controlled adaptive trial and open-label extension. Alzheimers Res Ther. 2016 Oct 18;8(1):44. doi: 10.1186/s13195-016-0210-1. PMID 27756421